CLINICAL TRIAL: NCT02098356
Title: Intradialytic Acid-base Changes and Organic Anion Production With High Versus Low Bicarbonate Hemodialysis
Brief Title: Comparison of High Versus Low Bicarbonate Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Matthew Abramowitz, Assistant Professor, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-480
Record Dates: First submitted 2014-03-24; First posted 2014-03-28 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-04

CONDITIONS: Chronic Kidney Disease; End-stage Renal Disease; Metabolic Acidosis
Keywords: hemodialysis; dialysis; acidosis; bicarbonate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low bicarbonate (Experimental): Low bicarbonate hemodialysis - 30 mEq/L dialysate bicarbonate
  Interventions: Other: Low Bicarbonate

INTERVENTIONS:
Other: Low Bicarbonate — Low bicarbonate hemodialysis - 30 mEq/L dialysate bicarbonate

SUMMARY:
This study will compare hemodialysis treatment with a standard, high-bicarbonate dialysis bath versus a lower bicarbonate dialysis bath, and will compare intradialytic acid-base changes and overall control of metabolic acidosis with the 2 treatment regimens.

DETAILED DESCRIPTION:
This study will compare hemodialysis treatment with a standard, high-bicarbonate dialysis bath versus a lower bicarbonate dialysis bath, and will compare intradialytic acid-base changes and overall control of metabolic acidosis with the 2 treatment regimens. These parameters will be assessed in patients currently receiving high-bicarbonate hemodialysis as part of usual care. They will then be switched to a lower bicarbonate prescription, after which these parameters will be reassessed. The study will also examine changes in inflammatory markers, glycemic control, ketogenesis, and lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Receiving chronic thrice-weekly conventional hemodialysis for at least 6 months

Exclusion Criteria:

* Use of oral alkali within the previous month
* Hospitalization within the previous month
* Inability to provide written informed consent
* Plans for kidney transplant in the next 2 months
* Planned change in phosphate binder therapy within the next month
* Pregnancy, or planned pregnancy in the next 2 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pre-dialysis serum bicarbonate | 5 weeks
  Change in predialysis bicarbonate

SECONDARY OUTCOMES:
serum beta-hydroxybutyrate | 5 weeks
  Change in beta-hydroxybutyrate during dialysis
beta-hydroxybutyrate clearance | 5 weeks
  Change in clearance between different dialysates
interleukin-6 | 5 weeks
  Change during dialysis
serum free fatty acids | 5 weeks
  Change during dialysis
Time to recover from dialysis | 5 weeks
  Change between dialysates
Dialysis symptom questionnaire | 5 weeks
  Change between dialysates

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abramowitz, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2014-05-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT02098356/ICF_000.pdf